CLINICAL TRIAL: NCT05705882
Title: China Nutrition Fundamental Data 2022
Acronym: CNFD 2022
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: National Institute of Hospital Administration, National Health Commission (Unknown)
Responsible Party: Principal Investigator, Wei Chen, Professor, Peking Union Medical College Hospital
Other Study IDs: I-22PJ744
Record Dates: First submitted 2023-01-12; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Nutritional Status of Chinese Inpatients; Nutritional Service Capacity of Medical Institutions in China

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Malnutrition — For the diagnosis of malnutrition, the investigators adopted the Global Leadership Initiative on Malnutrition (GLIM) scheme based on three phenotypic criteria (non-volitional weight loss, low body mass index, and reduced muscle mass) and two etiologic criteria (reduced food intake or assimilation, and inflammation or disease burden). To diagnose malnutrition at least one phenotypic criterion and one etiologic criterion should be present in patients with nutritional risk.

SUMMARY:
Malnutrition caused by reduced food intake or assimilation and varying degrees of acute or chronic inflammation is a serious and underappreciated risk factor for adverse clinical outcomes. Despite the substantial health and economic burden, malnutrition remains to affect a considerable proportion of hospitalized patients worldwide. Nationally representative studies from the USA, Australia, and European countries have reported prevalence figures in the range of 8.9% to 80.4%. However, national data in some resource-poor countries, such as China, the largest developing country in the world, are scarce.

During 2020 to 2022, the investigators conducted the China Nutrition Fundamental Data 2020 (CNFD 2020). This project provides a reference for nutritional risk assessment, malnutrition diagnosis, and treatment criteria for hospitalized patients in China. This project also provides data to promote the construction of clinical nutrition departments and improve the nutritional status of hospitalized patients. Thus, the investigators plan to conduct the China Nutrition Fundamental Data 2022 in a large, nationally representative sample of Chinese adult inpatients to 1) To further explore the relationship between nutrition and health; 2) To further understand the capacity of nutrition services in Chinese medical institutions.

This project will adopt a multistage, stratified, cluster-sampling procedure based on administrative divisions in China. For each participant, a structured interview will be done by trained nutritionists or clinicians. The following data will be acquired: weight change within and beyond six months, food intake change within two weeks, nutrition therapy during this hospitalization, Karnofsky score, clinical outcome, total hospitalization costs, and laboratory tests. The investigators will also collect information on participants' sociodemographic characteristics and medical history. The investigators will take physical measurements, including height, weight, waist circumference, hip circumference, mid-arm circumference, calf circumference, handgrip strength, and blood pressure following standard protocols. Body composition will be measured using bioimpedance analysis (BIA).

In addition, the investigators plan to collect information on the number of beds, the nutrition support team, the nutrition treatment plan and the construction of a full-time nutrition physician or nutrition nurse, the routine monitoring methods, interventions, and distribution of brochures for patients with malnutrition or nutritional risk in each project hospital.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Admitted to hospital within 24-48 hours (not emergency) due to tumor or digestive system, respiratory system, cardiovascular system, endocrine system, nervous system, and urinary system disease.

Exclusion Criteria:

* With mental illness or memory disorder who were unable to answer questions correctly
* Critically ill patients
* Lack behavioral ability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A large, nationally representative sample of Chinese adult inpatients
Sampling Method: Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of malnutrition | The day of the survey (day 1)
  For the diagnosis of malnutrition, the investigators adopted the Global Leadership Initiative on Malnutrition (GLIM) scheme based on three phenotypic criteria (non-volitional weight loss, low body mass index, and reduced muscle mass) and two etiologic criteria (reduced food intake or assimilation, and inflammation or disease burden). To diagnose malnutrition at least one phenotypic criterion and one etiologic criterion should be present in patients with nutritional risk.
Prevalence of nutritional risk | The day of the survey (day 1)
  Prevalence of nutritional risk was evaluated by Nutritional Risk Screening 2002 (NRS 2002). The minimum and maximum values were 0 and 7 respectively. Nutritional risk was defined as NRS 2002 score≥3. Higher scores mean higher nutritional risk.

CONTACTS AND LOCATIONS:
Locations (1):
- Dongcheng district，Peking union medical college hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided